CLINICAL TRIAL: NCT06804473
Title: Effect of Aerobic Exercise on Clinical Symptoms During the Ovarian Cycle
Acronym: OVARIANEXERCYC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Alberto Roldán, PhD, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OVARIANEXERCYCLE
Record Dates: First submitted 2025-01-21; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Primary Dysmenorrhea
Keywords: dysmenorrhea; exercise; pain; aerobic exercise
MeSH Terms: conditions — Dysmenorrhea; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The participants in the control group will continue with their usual care throughout the cycle without receiving the designed intervention. However, they will be asked to complete the follow-up questionnaires.
- Intervention group (Experimental): Participants in the experimental group will perform moderate-to-high intensity aerobic exercise on a stationary bicycle at the gym of Francisco de Vitoria University. The exercise intensity will range from 60-75% of their maximum heart rate (HRmax), with each session lasting 28 minutes, three times per week. The exercise protocol will involve interval aerobic training consisting of four intervals. Each interval will include:
  Warm up (5min) Active phase: 5 minutes at 60-75% HRmax, corresponding to a perceived exertion level of 5-7 on the modified Borg scale.
  Active recovery phase: 1 minute and 30 seconds at 30-50% HRmax, corresponding to a perceived exertion level of 2-3 on the modified Borg scale.
  Before starting the session, participants will complete a 5-minute warm-up on the stationary bicycle, progressively increasing intensity as follows: 3 minutes at 50-60% HRmax, 2 minutes at 60-70% HRmax Cool down (5min)
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — The exercise intensity will range from 60-75% of their maximum heart rate (HRmax), with each session lasting 28 minutes, three times per week. The exercise protocol will involve interval aerobic training consisting of four intervals
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effects of moderate-to-high intensity aerobic exercise on primary dysmenorrhea, a common condition characterized by painful menstrual cramps.

The study will involve women diagnosed with primary dysmenorrhea, who will be randomly assigned to one of two groups:

Experimental Group: Participants will perform a supervised aerobic exercise program tailored to their fitness level.

Control Group: Participants will continue their usual care without any additional interventions.

The study will run from February 2025 to April 2025 in Madrid, Spain. Before starting, all participants will complete a questionnaire to gather information about their demographics, menstrual cycle characteristics, medical history, and physical activity levels. This will help ensure an accurate diagnosis of primary dysmenorrhea and provide baseline data for comparison.

Participants will be randomly assigned to their groups using a computer-generated sequence, with allocation managed confidentially to avoid bias. The study's single-blind design ensures that the evaluators will not know the group assignments.

The goal of this research is to determine whether regular aerobic exercise can serve as an effective, non-pharmacological intervention to reduce the severity of menstrual pain and improve the quality of life for women with primary dysmenorrhea. The findings will inform patients, families, and healthcare providers about potential lifestyle strategies to manage this condition.

DETAILED DESCRIPTION:
This study investigates the potential benefits of aerobic exercise as a non-pharmacological intervention for primary dysmenorrhea, a condition that affects many women worldwide. Primary dysmenorrhea is characterized by painful cramps during menstruation without underlying pelvic pathology. It often disrupts daily life, leading to discomfort, reduced quality of life, and missed school or work days.

The study will be conducted in Madrid, Spain, between February 2025 and April 2025, and it involves women diagnosed with primary dysmenorrhea. Participants will be assigned to one of two groups using a randomized and single-blind design:

Experimental Group: Participants in this group will engage in a supervised aerobic exercise program tailored to their fitness level. The exercises will be moderate to high intensity, and they will follow established guidelines for safe and effective physical activity.

Control Group: Participants in this group will continue their usual care practices, such as using over-the-counter pain relievers, without additional interventions.

Study Procedures:

Eligible participants will first complete a comprehensive questionnaire. This form will gather key information, including demographic data, medical history, details about their menstrual cycles, and current physical activity levels. The diagnosis of primary dysmenorrhea will be confirmed based on clinical history, including characteristics of the pain, its onset with menstruation, accompanying symptoms, and the absence of indicators of secondary dysmenorrhea (e.g., irregular bleeding or unresponsiveness to NSAIDs).

Participants will be randomized in a 1:1 ratio using a computer-generated sequence, ensuring unbiased group assignment. An independent individual will manage the randomization process, and allocation will be concealed using sealed, opaque envelopes distributed sequentially as participants enroll in the study.

The primary goal is to evaluate whether regular aerobic exercise can reduce the severity of menstrual pain associated with primary dysmenorrhea. Secondary outcomes include assessing changes in quality of life, menstrual symptoms, and overall physical well-being.

Primary dysmenorrhea is commonly treated with medications such as nonsteroidal anti-inflammatory drugs (NSAIDs) or hormonal therapies. However, not all patients achieve relief, and some may prefer non-pharmacological approaches due to side effects or personal preferences. This study aims to explore aerobic exercise as a cost-effective, accessible, and safe alternative or complementary intervention.

The findings from this research may provide valuable insights for women seeking non-drug treatments for menstrual pain. If aerobic exercise proves effective, it could empower women with an evidence-based, proactive strategy to manage their symptoms. Healthcare providers may also gain additional tools to recommend as part of holistic care for patients with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria

* Age between 18 and 26 years.
* Sedentary lifestyle.
* Body Mass Index (BMI) between 18.5 and 26 kg/m².
* Regular menstrual cycle (24-38 days).
* Menstrual pain intensity ≥ 4 mm on the Visual Analog Scale (VAS).
* Presence of anxiety or stress.

Exclusion Criteria

* Pregnancy or breastfeeding within the last 3 months.
* Amenorrhea.
* Use of oral contraceptives in the last 3 months.
* Presence of an intrauterine device (IUD).
* Regular alcohol consumption.
* Active smoking.
* Chronic endocrine, digestive, neurological, or uncontrolled cardiovascular diseases, and/or psychiatric disorders.
* Any medical diagnosis contraindicating physical exercise.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 44 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain | Up to 8 weeks
  Menstrual pain intensity will be assessed using the Visual Analog Scale (VAS) 24 hours before the onset of menstruation and during menstruation. The scale ranges from 0 to 10, with higher scores indicating greater perceived pain intensity (Guillian, 2011). Participants will be required to complete the scale on menstrual days to evaluate their pain levels.

SECONDARY OUTCOMES:
Drug intake | Up to 8 weeks
  The use of analgesic medication will be recorded individually throughout the study to gather information on the amount consumed during the two menstruations evaluated during the intervention. This data will be analyzed to determine whether the designed exercise program influences the need for medication use (Armour, 2019).
Quality of life | Up to 8 weeks
  The participants' quality of life will be assessed using the SF-12 questionnaire, which consists of 12 questions with response options ranging from 3 to 5 points, depending on the question. Higher scores will indicate better health status. The questionnaire evaluates eight dimensions grouped into two main components: the physical component and the mental component (Schmidt, 2012; Ware, 1996).
Quality of life during menstrual bleeding | Up to 8 weeks
  Quality of life during menstrual bleeding days will be measured using the CVM-22 questionnaire, which comprises 22 questions evaluating the following components: health perception, physical and functional well-being, psychological and cognitive well-being, and menstrual-related symptoms. Higher scores on the CVM-22 indicate a worse quality of life during menstrual bleeding days (Pascual, 2019).
Sleep quality | Up to 8 weeks
  Sleep quality will be assessed using the Women's Health Initiative Insomnia Rating Scale (WHIIRS), which quantitatively evaluates the severity of insomnia. The scale consists of five questions assessing aspects such as difficulty falling asleep, nighttime awakenings, early morning awakenings, satisfaction with sleep, and daytime fatigue. Each question is scored from 0 (never) to 4 (always), yielding a global score ranging from 0 to 20 points, with a score above 9 indicating clinical relevance (Levine, 2003).
Stress, anxiety, and depression | Up to 8 weeks
  Stress, anxiety, and depression will be measured using the Depression, Anxiety, and Stress Scale - 21 (DASS-21). This self-report tool includes 21 statements and a 4-point response scale to assess experienced symptoms. Response options include: 0, "does not apply at all"; 1, "applies somewhat or occasionally"; 2, "applies to a considerable degree or often"; and 3, "applies very much or almost always." Higher scores on the DASS-21 indicate greater levels of depression, anxiety, or stress (Fonseca, 2010).
Adherence to the exercise program | Up to 8 weeks
  Adherence to the exercise program at Francisco de Vitoria University will be measured through attendance records for the sessions scheduled individually with each participant.

IPD SHARING:
Plan to Share IPD: Undecided
At this time, there are no plans to share individual participant data (IPD). The primary reason for this decision is to protect the confidentiality and privacy of participants, as sharing IPD may pose a risk of re-identification despite anonymization efforts. Additionally, the study does not have a specific framework or infrastructure in place for secure and compliant IPD sharing.
  However, summary data and results of the study will be disseminated through peer-reviewed publications and presentations at scientific conferences, ensuring that the scientific community and the public can benefit from the findings.

REFERENCES:
- [Background] Itani R, Soubra L, Karout S, Rahme D, Karout L, Khojah HMJ. Primary Dysmenorrhea: Pathophysiology, Diagnosis, and Treatment Updates. Korean J Fam Med. 2022 Mar;43(2):101-108. doi: 10.4082/kjfm.21.0103. Epub 2022 Mar 17. PMID 35320895